CLINICAL TRIAL: NCT06869044
Title: A Clinical Comparison of Two Soft Multifocal Contact Lenses - Proclear® 1 Day Multifocal and Clariti® 1 Day Multifocal 3 Add
Brief Title: A Clinical Comparison of Proclear® 1 Day Multifocal and Clariti® 1 Day Multifocal 3 Add
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-165
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Myopia; Hyperopia; Presbyopia
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- omafilcon A lenses first, then low ADD power somofilcon A lens (Experimental): Participants will wear two different types of study contact lenses, in a randomized order of testing for the two study contact lens types.
  Interventions: Device: omafilcon A lens; Device: Low ADD power somofilcon A lens
- omafilcon A lenses first, then medium ADD power somofilcon A lens (Experimental): Participants will wear two different types of study contact lenses, in a randomized order of testing for the two study contact lens types.
  Interventions: Device: omafilcon A lens; Device: Medium ADD power somofilcon A lens
- omafilcon A lenses first, then high ADD power somofilcon A lens (Experimental): Participants will wear two different types of study contact lenses, in a randomized order of testing for the two study contact lens types.
  Interventions: Device: omafilcon A lens; Device: High ADD power somofilcon A lens

INTERVENTIONS:
Device: omafilcon A lens — Participants will be randomized to wear omafilcon A lens for 15 minutes.
Device: Low ADD power somofilcon A lens — Participants will be randomized to wear low ADD power somofilcon A lens for 15 minutes.
  Arms: omafilcon A lenses first, then low ADD power somofilcon A lens
Device: Medium ADD power somofilcon A lens — Participants will be randomized to wear medium ADD power somofilcon A lens for 15 minutes.
  Arms: omafilcon A lenses first, then medium ADD power somofilcon A lens
Device: High ADD power somofilcon A lens — Participants will be randomized to wear high ADD power somofilcon A lens for 15 minutes.
  Arms: omafilcon A lenses first, then high ADD power somofilcon A lens

SUMMARY:
The aim of this study is to compare the overall lens satisfaction between two soft multifocal contact lenses.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the overall lens satisfaction between two soft multifocal contact lenses when compared to each other after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

1. They are at least 18 years of age.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They habitually use soft contact lenses (multifocal soft contact lenses, sphere lenses for monovision, sphere lenses for distance vision correction and spectacles for near vision correction,) and have done so for at least the past three months.
4. They have a minimum reading add of +0.75DS (based on their spectacle refraction)
5. They have spherical equivalent refractive error between +6.00 to -10.00DS at the corneal plane and refractive astigmatism of no greater than -0.75DC in each eye.
6. They are able to achieve distance HCVA of +0.10 logMAR or better in each eye.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are aphakic.
4. They have had corneal refractive surgery.
5. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall lens satisfaction | At the end of 15 minutes wear
  Overall Impression recorded on a visual analog scale of 0 to 100 where (0=Extremely poor. Unmanageable. Cannot use lenses, 100=Excellent. Highly impressed with these lenses overall.)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD, Ph.D, Principal Investigator — UC Berkeley
Locations (1):
- University of California, Berkeley, CA, Berkeley, California, United States